CLINICAL TRIAL: NCT03477097
Title: Frailty Prevention Through Improvement of Nutrition Physical Activity and Social Participation
Acronym: FPINPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Miaoli General Hospital, Ministry of Health and Welfare, Taiwan (Unknown)
Responsible Party: Principal Investigator, Wen-Harn Pan, Research Fellow, Academia Sinica, Taiwan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AS-IRB-BM-15020
Record Dates: First submitted 2016-01-11; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Frail Elderly
Keywords: Frailty; Social Determinants; Biological Risk Factors; Intervention; Cost Effectiveness
MeSH Terms: conditions — Frailty | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Control group w/o social network intervention (No Intervention): Subjects did not receive any intervention of nutrition, physical activity and social network.
- Control group w/ social network intervention (Experimental): Subjects only received the intervention of social network.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition group 1 w/o social network intervention (Experimental): Subjects only received the nutrition I intervention (e.g., food plate and multiple vitamin/ minerals powder).
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition group 1 w/ social network intervention (Experimental): Subjects received the nutrition I intervention (e.g., food plate and multiple vitamin/ minerals powder) and social network intervention as well.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition group 2 w/o social network intervention (Experimental): Subjects only received the nutrition II intervention (e.g., food plate, multiple vitamin/ minerals powder, fruit/vegetable concentrate capsule, and fish oil).
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition group 2 w/ social network intervention (Experimental): Subjects received the nutrition II intervention (e.g., food plate, multiple vitamin/ minerals powder, fruit/vegetable concentrate capsule, and fish oil) and social network intervention as well.
  Interventions: Other: Nutrition, exercise and social network intervention
- Physical activity group w/o social network intervention (Experimental): Subjects only received the personalized homed-based exercise prescription, which consisted of a combination of strength, flexibility, balance and endurance training.
  Interventions: Other: Nutrition, exercise and social network intervention
- Physical activity group w/ social network intervention (Experimental): Subjects received the personalized homed-based exercise prescription, which consisted of a combination of strength, flexibility, balance and endurance training, and social network intervention as well.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition 1 + physical activity group w/o social network (Experimental): Subjects received the nutrition I (e.g., food plate and multiple vitamin/ minerals powder) and exercise (e.g., personalized homed-based exercise plan) intervention.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition 1 + physical activity group w/ social network (Experimental): Subjects received the nutrition I (e.g., food plate and multiple vitamin/ minerals powder), exercise (e.g., personalized homed-based exercise plan), and social network intervention.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition 2 + physical activity group w/o social network (Experimental): Subjects only received the nutrition II (e.g., food plate, multiple vitamin/ minerals powder, fruit/vegetable concentrate capsule, and fish oil) and exercise (e.g., personalized homed-based exercise plan) intervention.
  Interventions: Other: Nutrition, exercise and social network intervention
- Nutrition 2 + physical activity group w/ social network (Experimental): Subjects only received the nutrition II (e.g., food plate, multiple vitamin/ minerals powder, fruit/vegetable concentrate capsule, and fish oil), exercise (e.g., personalized homed-based exercise plan), and social network intervention.
  Interventions: Other: Nutrition, exercise and social network intervention

INTERVENTIONS:
Other: Nutrition, exercise and social network intervention
  Arms: Control group w/ social network intervention; Nutrition 1 + physical activity group w/ social network; Nutrition 1 + physical activity group w/o social network; Nutrition 2 + physical activity group w/ social network; Nutrition 2 + physical activity group w/o social network; Nutrition group 1 w/ social network intervention; Nutrition group 1 w/o social network intervention; Nutrition group 2 w/ social network intervention; Nutrition group 2 w/o social network intervention; Physical activity group w/ social network intervention; Physical activity group w/o social network intervention

SUMMARY:
The life expectancy of the Taiwanese reached 75.98 years in males and 82.65 years in females in 2011. Because of the improved longevity and low birth rate, proportion of elderly population increased to 11.15% in our society. It is expected to be 21.2% in 2016. Frailty syndrome is an important path to disability or mortality in the elderly. Increase on disability will become a great burden to the society. This trend of population aging phenomenon occurs worldwide.

Frailty syndrome was defined by Fried el al. as older adults meet 3 of the following 5 conditions: (1) unintentional weight loss over 10 lbs in previous year, (2) weakness (grip strength at the lowest 20% by gender and BMI), (3) exhaustion (self-reported), (4) slowness (at the lowest 20% by gender and height), and (5) low physical activity. However, the definition of frailty is under discussion worldwide.

The sociological significance of frailty is that elders facing their changing roles in the society due to the changing position within the societal structure (i.e. moving from playing nuclear roles to marginal roles involuntarily or voluntarily) may potentially experience decline in psychosocial and physical well beings. Psychosocial and lifestyle factors and biomarkers are not well studied with respect to frailty. It is crucial to understand the social and biological risk factors of frailty and to design and study the possible prevention strategy for the prevention and management of frailty.

Therefore, the investigators propose to use randomization trials to investigate (1) the developmental process of frailty, the psycho-social determinants, related biomarkers and lifestyle factors; (2) the non-pharmaceutical intervention on preventing the progression of frailty and the cost-benefit of the intervention.

The investigators expect to (1) identify social determinants, biological and lifestyle factors which are associated with the development of frailty; (2) design and test clinical strategies to prevent frailty progression and (3) estimate the cost-effectiveness of the intervention. The results will have implications in public health education and in health policy making in order to prevent and to manage frailty in the elderly.

DETAILED DESCRIPTION:
This trial was conducted between October 2015 and June 2017 at the Miaoli General Hospital in Taiwan, and all eligible participants signed informed consent. The eligible pre-frail or frail elderly were screened according to the frailty phenotypes proposed by Fried and colleagues in the outpatient clinics. Participants who were over 65 years old and were able to walk 14 m independently were eligible for recruitment. The main exclusion criteria were critical illnesses; impairment in communication; nursing-home residents; participating other studies or taking nutritional supplementation; severe depression (Geriatric Depression Scale (GDS) < 10 points) or cognitive impairment (Mini Mental State Examination < 23 points). Participants were randomly assigned into study groups for 3-month intervention and 3-month self-maintenance period. The assessment of all participants were conducted by blind case managers at baseline, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* To walk 14 meters within 1 minute by him-/ her-self
* Fried score is in the range of 1 to 5 points
* To be willing to join 3-month intervention

Exclusion Criteria:

* Having sever disease (i.e., cancer, under intensive care, or survival time < 6 months)
* Having communication problem (i.e., hearing-impaired, visually disabled, aphasia, dementia, or schizophrenia)
* Stay in the nursing home or other similar institutes
* Having joined other study
* Not willing to take the food supplement of multiple vitamin, fruit/vegetable concentrate capsule, and fish oil
* GDS > = 10 points or MMSE < 24 (If he/ she is illiteracy, MMSE < 17)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Frailty score (Score range: 0-5, higher scores indicate worse performance) | 6 months
  Based on the Cardiovascular Health Study criteria, the frailty phenotypes were quantified by frailty score, which was the primary outcome in this study.

SECONDARY OUTCOMES:
Handgrip strength | 6 months
  Physical performance measure
Gait speed | 6 months
  Physical performance measure
Back scratch | 6 months
  Physical performance measure
Sit and reach | 6 months
  Physical performance measure
Standing heel-rise | 6 months
  Physical performance measure
Geriatric Depression Scale (Score range: 0-15, higher scores indicate worse performance) | 6 months
  Mental Health measure
Mini Mental State Examination (Score range: 0-30, higher scores indicate better performance) | 6 months
  Mental Health measure
Short form-12 mental component summary score (Score range: 0-100, higher scores indicate better performance) | 6 months
  Mental Health measure

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica
Locations (1):
- Miaoli General Hospital, Miaoli, Taiwan

REFERENCES:
- [Derived] Hsieh TJ, Su SC, Chen CW, Kang YW, Hu MH, Hsu LL, Wu SY, Chen L, Chang HY, Chuang SY, Pan WH, Hsu CC. Individualized home-based exercise and nutrition interventions improve frailty in older adults: a randomized controlled trial. Int J Behav Nutr Phys Act. 2019 Dec 2;16(1):119. doi: 10.1186/s12966-019-0855-9. PMID 31791364